CLINICAL TRIAL: NCT02837302
Title: Branched-chain Amino Acid (BCAA) on Progression of Advanced Liver Disease (BRAVE): Korean Nation-wide Multicenter Retrospective and Prospective Observational Cohort Study
Brief Title: Branched-chain Amino Acid (BCAA) on Progression of Advanced Liver Disease
Acronym: BRAVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Samil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Won Young Tak, Division of Gastroenterology & Hepatology, Kyungpook National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAVE_prospective
Record Dates: First submitted 2014-05-13; First posted 2016-07-19 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Liver Cirrhosis
Keywords: Liver cirrhosis; Branched chain amino acid; End-Stage Liver Disease score
MeSH Terms: conditions — Liver Cirrhosis | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Livact (Active Comparator): Daily dose of 12.45g of branched-chain amino acid containing 3.4g of L-valine, 5.7g of L-leucine, and 2.9g of L-isoleucine over 6 months.
  Interventions: Drug: Livact
- General nutritional support (No Intervention): General nutritional support

INTERVENTIONS:
Drug: Livact — Daily dose of 12.45g of branched-chain amino acid containing 3.4g of L-valine, 5.7g of L-leucine, and 2.9g of L-isoleucine over 6 months.
  Other Names: Branched chain amino acid
  Arms: Livact

SUMMARY:
Protein-calorie malnutrition is frequently observed in patients with advanced liver cirrhosis. There have been continued interests in potential benefits of long-term oral branched-chain amino acid supplement in improving severity of liver disease. However, there are limited evidences in literature. The aim of this study is to evaluate the efficacy of oral branched-chain amino acid in patients with advanced liver cirrhosis.

DETAILED DESCRIPTION:
This study is a multicenter retrospective cohort study involving thirteen centers in Korea nation-wide. The inclusion criteria are liver cirrhosis patients with Child-Pugh score 8 to 10. The major exclusion criteria are abnormal serum creatinine level, and hepatocellular carcinoma with viable tumor. The investigators analyzed improvement of Model for End-Stage Liver Disease score, Child-Pugh score, incidence of cirrhosis-related complications, and event free survival.

ELIGIBILITY:
Inclusion Criteria:

* Advanced liver cirrhosis patients with Child-Pugh score 8 to 10

Exclusion Criteria:

* Diagnosis of malignancy (except hepatocellular carcinoma) within 3 years or untreated malignancy
* Major organ failure (heart, lung and kidney) need to admission or medical therapy or dialysis
* Patients already on a waiting list or being considered for major organ transplantation.
* Serum creatinine above upper normal range (>1.5 mg/dL)
* Patients treating with albumin replacement regularly
* Viable hepatocellular carcinoma or advanced Barcelona Clinic Liver Cancer stage or hepatocellular carcinoma below 6 months life expectancy
* Patients being impossible to secession of alcohol consumption
* Patients being impossible to oral ingestion or oral medication
* Pregnancy or being considered for pregnancy
* Breast feeding
* Amyotrophic lateral sclerosis
* Patients with other metabolic disorder presenting branched-chain ketoaciduria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1470 (Estimated)
Dates: Start 2012-11; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
End-Stage Liver Disease score was calculated using serum total bilirubin, creatinine, international normalized ratio | After enrollment, the patients was assessed every 3 or 6 months for 2 years or until death

SECONDARY OUTCOMES:
Incidence of cirrhosis-related complications including death | After enrollment, the patients was assessed every 3 or 6 months for 2 years or until death

CONTACTS AND LOCATIONS:
Overall Officials: Won Young Tak, M.D., Ph.D., Principal Investigator — Kyungpook national university hospital, department of internal medicine
Locations (1):
- Kyungpook national university hospital, Daegu, South Korea